CLINICAL TRIAL: NCT05470543
Title: Effect of Nurse-led Supportive Care on Caregiver Burden and Well-being Among Primary Caregivers of Women With Breast Cancer: A Pragmatic Parallel Group Randomized Controlled Trial
Brief Title: Effect of Nurse-led Supportive Care on Caregiver Burden and Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Pinar Zorba Bahceli, PhD RN, Assistant Professor, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019/639
Record Dates: First submitted 2022-07-19; First posted 2022-07-22 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Nurse-led Supportive Care
Keywords: Breast cancer; Caregiver burden; Well-being; Nurse-led care
MeSH Terms: conditions — Breast Neoplasms; Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-led Supportive Care Group (Experimental)
  Interventions: Behavioral: Nurse-led supportive care
- Control Group (No Intervention): The control group received only usual care. They did not receive any intervention during the study period.

INTERVENTIONS:
Behavioral: Nurse-led supportive care — Nurse-led supportive care was given to primary caregivers of women with breast cancer. Nurse-led supportive care was applied to primary caregivers for eight weeks in the form of face-to-face clinic interviews. It took an average of 30 minutes to interview with primary caregivers at the clinic.
  Arms: Nurse-led Supportive Care Group

SUMMARY:
Breast cancer is the most common type of cancer in women with a high mortality rate in the world. Women may experience many different physiological and psychological symptoms (such as pain, nausea-vomiting, fatigue, stress, anger, and isolation) during diagnosis and treatment process. Family members often become caregivers at the time of diagnosis, and treatment of breast cancer patients. Therefore, family caregivers experience burden and poor health-related quality of life.

DETAILED DESCRIPTION:
This a pragmatic, parallel group randomized controlled trial aimed that investigating the effect of nurse-led supportive care on caregiver burden and well-being among primary caregivers of women with breast cancer. This trial was conducted in the chemotherapy outpatient clinic of training and research hospital located in Turkey. All primary caregivers were family members.

ELIGIBILITY:
Inclusion Criteria:

* Being the primary caregiver of breast cancer patients
* Literate
* Able to understand and complete the questionnaires
* Willingness to participate in the study

Exclusion Criteria:

* Having communication problems
* Having psychological diseases
* Receiving any supportive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2022-12-24 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Zarit Burden Interview (ZBI) | Change from baseline Zarit Burden Interview score at 9th weeks.
  The ZBI is a measure of caregiving burden developed by Zarit et al. (1980). The Turkish version of this scale has been validated by Inci and Erdem (2018). It consists of 22 items, and responses are recorded on a five-point Likert scale. The level of caregiver burden can be ascertained based on the total scale scores, which range from 0 to 88. Higher scores indicate a higher level of caregiver burden.The Cronbach's α of the Turkish version of this scale was 0.91 in Inci and Erdem (2018) validation study

SECONDARY OUTCOMES:
Caregiver Well-Being Scale | Change from baseline Caregiver Well-Being Scale score at 9th weeks.
  The scale was developed by Berg-Weber et al. (2000) in order to measure the level of caregivers of patients with chronic diseases to meet their basic needs and activities of living. The scale is made up of two subscales, namely, basic needs and activities of living, which try to measure the daily activity level of the caregivers. It consists of 44 items, and responses are recorded on a five-point Likert scale. Higher scores indicate a higher level of well-being. The Cronbach's α of the Turkish version of this scale was 0.86 in Demirtepe and Bozo (2009) validation study.

CONTACTS AND LOCATIONS:
Overall Officials: Pinar Zorba Bahceli, PhD, Principal Investigator — Izmir Bakircay University Faculty of Health Sciences Izmir, Turkey, 35560
Locations (1):
- Izmir Bakircay University Faculty of Health Sciences, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No